CLINICAL TRIAL: NCT07201805
Title: Effects of Early Physiotherapy on Motor Optimality Score in At-Risk of Infants: A Double-Blind Randomized Controlled Study
Brief Title: Effects of Early Physiotherapy on Motor Optimality Score in At-Risk of Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate profesor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Early PT on Motor Optimality
Record Dates: First submitted 2025-09-15; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Infants Admitted to Neonatal Units; Preterm; Physiotherapy and Rehabilitation; Family Centered
MeSH Terms: conditions — Premature Birth | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Physiotherapy Program (Experimental): A physiotherapy program tailored to the needs of infants from families who volunteer to participate will be implemented until and with family recommendations at the time of discharge. Parents of all at-risk infants will receive advice on handling, carrying, and positioning at the time of discharge.
  Interventions: Other: Early Physiotherapy Program
- Standard of care (Other): Babies from families unable to attend physiotherapy for any reason (working parents, those unable to attend treatment sessions, or those living out of town) will constitute the control group, provided they are available for evaluation. The control group will receive routine developmental NICU care, as well as one-time instruction in positioning and holding and carrying principles upon discharge.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Early Physiotherapy Program — The physiotherapy program provided upon discharge will consist of family education programs that include parental contact and therapeutic holding, carrying, positioning, and sucking facilitation to stimulate postural responses. The physiotherapist will provide training to integrate these programs into daily routines. The physiotherapy group will receive a routine-based family collaborative early intervention program. This program will consist of family education programs based on a goal-oriented model of active motor learning and sensory strategy development for the baby in an enriched environment, incorporating holding, carrying, and positioning into daily routines. If possible, the entire family will participate in these programs.
  Arms: Early Physiotherapy Program
Other: Control group — The control group will be shown one-time positioning and holding and carrying principles in addition to routine developmental NICU care at the time of discharge.
  Arms: Standard of care

SUMMARY:
Medical and technological advances in neonatal care have led to a decrease in neonatal mortality and an increase in the survival of very low birth weight infants, leading to a global increase in the prevalence of cerebral palsy (CP), cardiorespiratory disorders, blindness, cognitive delays, and hearing impairments. Early diagnosis and intervention programs have been established to meet the developmental needs of these at-risk infants in the neonatal intensive care unit (NICU). The goal of these programs is to facilitate the development of at-risk infants and normalize their motor, cognitive, and sensory development.Research remains unclear about which interventions are more effective when implemented. It is known that early intervention improves motor development in these infants, and that programs that include parents have more positive long-term outcomes for the cognitive and language development of at-risk infants.General Movements (GMs) are spontaneous movements that occur from the fetal period to 18 weeks postterm. Prechtl's General Movements Assessment (GMA) is a reliable tool for functional assessment of the young central nervous system.The assessment of motor repertoire (via the motor optimality score, MOS) describes the quality and quantity of the concurrent motor repertoire recorded during the GM assessment.The revised motor optimality score (MOS-R) has the potential to increase the prediction of adverse neurodevelopmental outcomes. It is noteworthy that the literature contains limited studies examining the effect of early physiotherapy applied to at-risk infants after NICU discharge on MOS-R. Therefore, the aim of this planned study was to investigate the effect of early family collaborative physiotherapy approaches applied to at-risk infants after NICU discharge on GMs MOS-R. Another aim was to determine the effect of early physiotherapy on neurological examination, cognitive, and language development in infants at 3 and 6 months of age and to compare them with similar peers receiving a routine treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with periventricular hemorrhage (PVH), intracranial hemorrhage (ICH), cystic PVL, HIE, kernicterus, perinatal asphyxia, neonatal sepsis, necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), RDS, or BPD, and those receiving oxygen or mechanical ventilation (MV) support
* Infants with a 5-minute Apgar score <3, <37 weeks' gestation, <1500 grams of preterm birth, or prematurity due to multiple births.
* Infants with the corrected age of 2 to 4 months

Exclusion Criteria:

* Infants with congenital malformations (spina bifida, congenital muscular torticollis, arthrogryposis multiplex congenita, etc.), babies diagnosed with metabolic and genetic diseases (down syndrome, spinal muscular atrophy, duchenne muscular dystrophy, etc.)

Ages: 2 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Motor Optimality Score for 3-to 5-Month-Old Infants - Revised and Motor Repertoire Score | postterm 12th to 20 weeks of age
  All babies will have their Motor Optimality Scores (MOS-R) calculated at the end of the 4th and 5th months, adjusted for fidgety General Movements of the videos. The MOS-R assesses movement repertoire and scores in the following four areas.The total of these scores varies between 5 and 28. Higher scores shows better developmental status.
Pretchl's General Movements (GMs) Assesment | after the postterm 8th weeks of age and after the postterm weeks of 12 to 20 weeks
  General movements (GMs) are the spontaneous repertoire of movements present from early fetal life until the 20th week postpartum. They are writhing until the 8th week postpartum and then fidgety until approximately the 20th week.Video recordings will begin in the NICU three days after birth in the preterm period. All infants will be examined for writhing and fidgety movements (FM) via video recordings.Movements during the preterm and writhing periods will be classified as PR, CS, and Ch GMs or normal. Movements during the fidgety period will be recorded as F+ or F++ when normal, AF when abnormal, or F- when not observed.

SECONDARY OUTCOMES:
Hammersmith Neonatal Neurological Examination (HNNE) | from birth to 42 weeks of age
  This measurement has been developed by Dubowitz, the examination standardized optimality scores by evaluating low-risk term and high-risk preterm infants at term age. The scale consists of a 34-item proforma. This proforma includes tone (10), tone patterns (5), reflexes (6), movements (3), abnormal signs (3), and behavior (7). All items are scored from 1 to 3 (half points are also possible). Higher scores indicate better neurological status.
Hammersmith Infant Neurological Examination (HINE) | 2th, 3th, 6th months of corrected age
  The Hammersmith Infant Neurological Examination (HINE) is a simple, standardized, and scoreable test for the clinical neurological assessment of infants aged 2-24 months. HINE consists of a total of 37 items, divided into three sections: neurological examination, developmental motor milestones, and behavioral status.It consists of three sections: (1) a neurological examination that assesses cranial nerve function, posture, movements, tone, reflexes, and reactions; (2) motor milestones; and (3) behavior. Each of the 26 items on the test is initially scored individually (0, 1, 2, 3, or half points). A total score is then calculated, with miimum score of 37 and a maximum score of 78 points.A higher score indicates better neurological status.
BAYLEY-III Infant and Child Development Assessment Scale (BAYLEY-III) | 3th and 6th months of corrected age
  The BAYLEY-III Infant and Child Development Assessment Scale (BAYLEY-III ) is a neurocognitive assessment used to monitor the development of infants aged 0-42 months. It comprises five domains: cognitive, language, motor, social-emotional, and adaptive functions. This study will assess only the cognitive, language, and motor domains.To ensure comparability of results from the 5 domains, a composite score is calculated for each domain (mean 100±15). A composite score below 2 standard deviations (SD) (<70) is considered a severe delay across all domains.Higher scores give better developmental stages.
Sociodemographic form | baseline
  Sociodemographic information and prenatal/perinatal risks (MRI, cUS results, diagnosis, neurological evaluation) of all infants and their parents will be obtained from hospital records after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubet, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No